CLINICAL TRIAL: NCT02784847
Title: A Pilot Trial of Triheptanoin for the Preventive Treatment of Migraine
Acronym: TRIMI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX007
Record Dates: First submitted 2016-03-10; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment arm (Other): pilot-study with single arm of 10 migraine patients treated for 3 months with triheptanoin 1mg/kg/day
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin oil administered three times per day during meals at a total dose 1mg/kg/day for 3 months
  Other Names: UX007

SUMMARY:
A pilot trial of triheptanoin, a natural compound able to promote anaplerotic mitochondrial metabolism, for the preventative treatment of migraine.

DETAILED DESCRIPTION:
To test the ability of a daily 3-month treatment with triheptanoin to prevent migraine attacks in 10 migraine patients.

This is an open, non-randomized pilot trial that might justify a placebo-controlled trial, if there are at least 50% of patients with ≥50% reduction in attack frequency.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-65 years old having an effective contraception or being menopaused
* Diagnosis of migraine without aura (ICHD3beta 1.1) since at least 2 years
* 4-10 migraine days per month during the last 3 months
* No preventive anti-migraine therapy during the last month

Exclusion Criteria:

* > 4 tension-type headache episodes per month
* Medication overuse headache or other headache types
* Resistance to >3 previous preventive anti-migraine drug treatments
* Any serious medical or psychiatric condition
* On-going or previous bowel disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change in monthly migraine days | Between the 1-month baseline and the 3rd month of triheptanoin treatment

SECONDARY OUTCOMES:
Change in mean attack severity | Between the 1-month baseline and the 3rd month of triheptanoin treatment
Change in mean attack duration | Between the 1-month baseline and the 3rd month of triheptanoin treatment
Number of patients who have at least a 50% reduction in monthly migraine days | Between the 1-month baseline and the 3rd month of triheptanoin treatment

OTHER OUTCOMES:
Tolerance and gastrointestinal adverse effects | During the 3 months of triheptanoin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schoenen, MD,PhD, Principal Investigator — University Hospital Liège

IPD SHARING:
Plan to Share IPD: No